CLINICAL TRIAL: NCT05058118
Title: A Randomized, Double-Blind, Single-Dose, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of FL058 for Injection in Healthy Chinese Subjects.
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of Intravenous FL058 Administered in Healthy Subjects(SAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FL058-I-01
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FL058 (Experimental): a single ascending dose (SAD) of intravenous (IV) FL058(50mg~2000mg)
  Interventions: Drug: FL058
- Placebo (Placebo Comparator): FL058 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FL058 — 50mg、250mg、500mg、1000mg、1500mg、2000mg
  Arms: FL058
Drug: Placebo — empty bottle
  Arms: Placebo

SUMMARY:
To evaluate the safety,tolerability and pharmacokinetics of single intravenous doses of FL058 in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 18 and 45 years (inclusive).
2. Body mass index (BMI) ranges from 19 to 26 kg/m2 (inclusive), and the body weight is ≥50kg.
3. Good general health as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory tests.
4. Provide voluntary written informed consent prior to any study procedures and are willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

1. Concurrent or history of clinically significant cardiovascular, hepatic, renal, endocrine, gastrointestinal, respiratory, psychiatric, neurologic and/or hematological disorders.
2. Positive screen result for HBsAg, HCV-Ab, or HIV-Ab at screening.
3. History of clinically significant food or drug allergy.
4. A QT interval corrected using Fridericia's formula >450 msec.
5. eGFR<90mL/min/1.73m2.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events [Safety and Tolerability] | Day 1 to Day 7

SECONDARY OUTCOMES:
FL058 -Cmax | Up to 48 hours post-dose
  To evaluate the PK of single intravenous doses of FL058 in healthy adult human subjects.
FL058 -AUC | Up to 48 hours post-dose
  To evaluate the PK of single intravenous doses of FL058 in healthy adult human subjects.
FL058 -t1/2 | Up to 48 hours post-dose
  To evaluate the PK of single intravenous doses of FL058 in healthy adult human subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, China

REFERENCES:
- [Derived] Huang Z, Yang X, Jin Y, Yu J, Cao G, Wang J, Hu Y, Dai J, Wu J, Wei Q, Tian Y, Yu S, Zhu X, Mao X, Liu W, Liang H, Zheng S, Ju Y, Wang Z, Zhang J, Wu X. First-in-human study to evaluate the safety, tolerability, and population pharmacokinetic/pharmacodynamic target attainment analysis of FL058 alone and in combination with meropenem in healthy subjects. Antimicrob Agents Chemother. 2024 Jan 10;68(1):e0133023. doi: 10.1128/aac.01330-23. Epub 2023 Dec 6. PMID 38054726